CLINICAL TRIAL: NCT00965640
Title: A Prospective, Single Center, Open Label, Proof of Principle Study to Assess the Efficacy and Safety of 150 Units of Botulinum Toxin-A Intra-Muscular Injection in the Prevention of Hair Loss in Men With Androgenetic Alopecia
Brief Title: Treatment of Male Pattern Baldness With Botulinum Toxin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Crown Institute (Other)
Responsible Party: Dr. B. Freund, Principal Investigator, Crown Institute
Purpose: Screening
Other Study IDs: MPB-2002-01; HPB 081023
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Male Pattern Baldness
Keywords: male pattern baldness; androgenetic alopecia; hair loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botulinum Toxin - A injections

SUMMARY:
This proof of concept study seeks to demonstrate that Botulinum toxin injections are a safe and effective method for treating this form of hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Male pattern baldness
* Norwood II-VI

Exclusion Criteria:

* Treatment with Botulinum toxins or other hair growth interventions with past year

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2002-12; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Hair Growth | 1 year

SECONDARY OUTCOMES:
Hair Loss | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brian Freund, MD, Principal Investigator — Crown Institute
Locations (1):
- Crown Institute, Pickering, Ontario, Canada

REFERENCES:
- [Derived] Freund BJ, Schwartz M. Treatment of male pattern baldness with botulinum toxin: a pilot study. Plast Reconstr Surg. 2010 Nov;126(5):246e-248e. doi: 10.1097/PRS.0b013e3181ef816d. No abstract available. PMID 21042071